CLINICAL TRIAL: NCT06505811
Title: City of Pomona's Guaranteed Income Program for Parents With Children Under the Age of Give
Brief Title: Mixed Methods Evaluation of the Pomona Household Universal Grant (HUG) Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Conrad N. Hilton Foundation (Other); City of Pomona (Unknown); FORWARD Platform (Unknown)
Responsible Party: Principal Investigator, Judith L. Perrigo, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 23-001551
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Early Child Well-being; Parental Stress; Family Economic Security; Parental/Caregiver Health; Mental Health
Keywords: early child development; guaranteed Income; unconditional cash transfer; parent-child relationship; poverty; financial security
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: All eligible applicants will be entered into a lottery which will randomly select a total of 600 participants for the Pomona Household Universal Grant (HUG) program. Selected applicants will be assigned to one of the following groups (July 2024):
  Treatment Group - 250 applicants will receive 18 monthly payments in the amount of $500 each Control Group - 350 applicants will receive $20 stipend payments for a total of 18 months
Who Masked: Participant, Outcomes Assessor
Masking Description: The assessors completing the in-home observations will not be apprised of treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treated Group ($500 GI for 18 months) (Experimental): Treated Group will receive $500 per month for 18 months (anticipated n=250)
  Interventions: Behavioral: Guaranteed Income ($500/monthly)
- Comparison Group ($20 GI for 18 months) (Active Comparator): Comparison Group will receive $20 per month for 18 months (anticipated n=350)
  Interventions: Behavioral: Active Comparison ($20/monthly)

INTERVENTIONS:
Behavioral: Guaranteed Income ($500/monthly) — Participants receive $500 monthly for up to 18 months.
  Arms: Treated Group ($500 GI for 18 months)
Behavioral: Active Comparison ($20/monthly) — Participants receive $20 monthly for up to 18 months.
  Arms: Comparison Group ($20 GI for 18 months)

SUMMARY:
The City of Pomona is launching the Pomona Household Universal Grant (HUG) program in the Summer of 2024. Pomona HUG is a pilot project that will provide 250 parents/caregivers with children under 5 years old $500 a month for 18 months. Pomona's guaranteed income (GI) initiative provides relief for the most economically vulnerable households. The study will investigate the impacts of GI on financial security, material hardship, health and well-being, food security, social support, parenting, and childhood development. The intervention group will be compared to a control group of 350 parents/caregivers receiving only a nominal ($20) amount per month during the 18 month period.

DETAILED DESCRIPTION:
GI programs are commonly depicted as catalysts for reshaping social welfare paradigms. Such programs not only address immediate material hardship through consistent and unconditional financial support but also have the potential to confer broader societal benefits. For instance, GI programs can reduce income inequality, enhance socio-economic conditions, and improve health outcomes and overall well being.

The early years of a child's life hold profound significance, as approximately 90% of brain development occurs before age five. This period lays the crucial foundation for lasting effects, presenting a valuable opportunity to implement an innovative, two-generation GI initiative in Pomona, California. By adopting a comprehensive two-generation approach, Pomona can pave the way for transformative change in equipping parents/caregivers with the means to secure basic necessities such as food, clothing, and shelter for themselves and their children. By alleviating the stress of financial instability, parents/caregivers are empowered to focus on their education, skill development, career prospects, and responsive parenting. Consequently, the ripple effects hold promise to disrupt the cycle of poverty, offering a brighter future for both children and their families.

The investigators guiding research questions are to examine how GI impacts child, parent/caregiver, and family outcomes. The evaluation utilizes a mixed methods approach, employing a randomized controlled trial (RCT) design which includes parent surveys, home-based observations, and semi-structured qualitative interviews.The study includes a total of N=600 dyads (parent/caregiver and child), with n=250 receiving $500 GI monthly for 18 months and a control group of n=350 receiving $20 per month for the same duration. Baseline, and follow-up surveys at year 1 and year 2 will be administered to all participants. Home observations will be conducted with all 600 participants to better understand the impact of GI on parent-child relationships. Lastly, qualitative interviews will be conducted with a subset of parents receiving GI (n=30) and those who do not (n=30) to gain a deeper understanding of the intervention's impact.

ELIGIBILITY:
Inclusion Criteria:

Must live in the City of Pomona;

Must be 18 years old upon application submission;

Must be the parent or legal guardian of a child aged prenatal to under 4 years old at the time of application;

Must meet at least one of the following qualifiers (#1-4):

Experienced negative impact due to the Covid-19 pandemic including:

* The participant or anyone in the participant's household experienced unemployment during the pandemic.
* The participant or anyone in the participant's household experienced increased food or housing insecurity during or as a result of the pandemic.

Home address is located within a qualified census tract (QCT).

Participant currently receiving any of the below benefits:

* Federal Pell Grants
* Free-and Reduced-Priced Lunch (NSLP) and/or School Breakfast (SBP) programs
* Head Start and/or Early Head Start
* Low Income Housing Energy Assistance Program (LIHEAP)
* Section 8 Vouchers : Public Housing & Housing Choice Vouchers
* Supplemental Security Income (SSI) - Social Security
* CalFresh or SNAP (Supplemental Nutrition Assistance Program)
* Temporary Assistance for Needy Families (TANF)
* Supplemental Nutrition Program for Women, Infants, and Children (WIC)
* Medicaid or MediCal
* Children's Health Insurance Program (CHIP)
* Childcare Subsidies through Child Care Development Fund (CCDF) Program
* Household income is at or below 65% AMI (Area Median Income)

In order to be approved for the program, the participant agrees to Informed Research Consent.

Exclusion Criteria:

Individuals that do not meet one or more of the inclusion criteria listed above.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Financial Security | Measured at baseline, 1-year after the start of the intervention, and at follow-up (6 months post-intervention period)
  Investigators use the Financial Well-being Scale developed and tested by the Consumer Financial Protection Bureau. Raw totals are derived from the participant responses which is then converted to a financial well-being score. Scores for the self-administered abbreviated version of the scale range from 19-90. Higher scores represent a higher level of reported financial well-being.
Early Childhood Well-being | Measured at baseline, 1-year after the start of the intervention, and at follow-up (6 months post-intervention period)
  Investigators use the developmental milestones subdomain from the Survey of Well-being of Young Children (SWYC) to measure early childhood well-being. The SWYC milestones subdomain assesses the cognitive, language, and motor development of children. Respondents are asked a set of 10 questions based on their child's age. Responses are scored and total scores range from 0 - 20. A cut off is provided for each age group and when the score is above this cutoff, it indicates that a child appears to be meeting age expectations for development.

SECONDARY OUTCOMES:
Parent-child interactions | Measured at baseline, 1-year after the start of the intervention, and at follow-up (6 months post-intervention period)
  Investigators measure this using the Healthy Families Parenting Inventory (HPFI) - Subdomain: Parent/Child Interaction, comprised of 10 questions. Reverse scoring is implemented for a set of questions. Total scores range from 10-50.
Food security | Measured at baseline, 1-year after the start of the intervention, and at follow-up (6 months post-intervention period)
  Investigators use the six-item short form of the United States Department of Agriculture Food Security Survey Module. Total scores range from 0-6 with higher scores indicating increased levels of food insecurity.
Parent/caregiver stress | Measured at baseline, 1-year after the start of the intervention, and at follow-up (6 months post-intervention period)
  Investigators use the Parental Stress Scale to measure parent/caregiver stress. Scores from the Parents Stress Scale range from 18-90. Before summing participant scores, reverse scoring is implemented for several items. Higher scores represent higher levels of parental stress.

CONTACTS AND LOCATIONS:
Overall Officials: Judith L Perrigo, PhD, Principal Investigator — University of California, Los Angeles; Daniel Eisenberg, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant survey data and home observation data will be available upon request and completion of a data access agreement. The deidentified data will be available to investigators with a proposal approved by an Institutional Review Board (or other independent review committee).
Supporting Information: Study Protocol, ICF
Time Frame: Proposals may be submitted for PI review 6 months following publication of the study's primary results (which is estimated to be 1-2 years following project completion). The PI will review such requests for up to 5 years after such publication.
Access Criteria: Proposals should be directed to Dr. Judith Perrigo at jperrigo@luskin.ucla.edu.

REFERENCES:
- [Background] Krysik J, Lecroy CW. Development and initial validation of an outcome measure for home visitation: The healthy families parenting inventory. Infant Ment Health J. 2012 Sep;33(5):496-505. doi: 10.1002/imhj.21343. Epub 2012 Jun 15. PMID 28520271
- [Background] Berry, J. O., & Jones, W. H. (1995). The parental stress scale: Initial psychometric evidence. Journal of social and personal relationships, 12(3), 463-472.
- [Background] Perrin, E. C., Sheldrick, R. C., Visco, Z., & Mattern, K. (2016). The survey of well-being of young children (SWYC) user's manual. Boston, MA: Floating Hospital for Children at Tufts Medical Center.
- [Background] Call CC, Boness CL, Cargas S, Coakley KE. Measuring food security in university students: A comparison of the USDA 10-item and six-item food security survey modules. J Hunger Environ Nutr. 2024;19(6):1325-1342. doi: 10.1080/19320248.2024.2310485. Epub 2024 Jan 30. PMID 39735215
- [Background] Consumer Financial Protection Bureau (CFPB). Measuring financial well-being: A guide to using the CFPB Financial Well-Being Scale. 2015.